CLINICAL TRIAL: NCT01522274
Title: Efficacy of Brisk Walking as a Smoking Cessation Treatment Adjunct Among Women
Brief Title: Quit Smoking With Nicotine Patch and Exercise/Health Education (Females Only)
Acronym: QFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David M. Williams, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CA155381; R01CA155381 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate intensity exercise (Active Comparator): Brisk walk on treadmill for 56 minutes 3x per week.
  Interventions: Behavioral: Moderate intensity exercise
- Health education (Active Comparator): Attend health education sessions 3x per week.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Moderate intensity exercise — Brisk walking on a treadmill for 56 minutes 3x per week.
  Arms: Moderate intensity exercise
Behavioral: Health education — Videos
  Arms: Health education

SUMMARY:
This research study is for FEMALE cigarette smokers who want to quit smoking.

Participants will be provided with brief quit-smoking education at the beginning of the study and will receive the nicotine patch for 10 weeks, free of charge.

Participants will be assigned to either an exercise program or a general health education program. The exercise and health education programs will take place over 14 weeks, with follow-up appointments 3, 6, and 12 months after the end of the 14-week program.

There is no fee for any part of this study and participants will be compensated for their time.

DETAILED DESCRIPTION:
Participants must complete telephone screening process first.

All eligible participants must attend an orientation session when the investigators will explain the study in detail. After this session, interested participants will complete a consent form and the investigators will collect blood pressure, resting heart rate, body mass index (height/weight), and a carbon monoxide sample to confirm eligibility. The investigators will then explain the physician consent process (all eligible and interested participants must obtain consent from a physician or clinic that they have seen in the past year to confirm that it is safe for them to participate).

ELIGIBILITY:
Inclusion Criteria:

* Current smoker

Exclusion Criteria:

* Ineligible after telephone screen.
* Each participant's personal physician/clinic determines it is unsafe to participate.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2012-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | 7-Day Point Prevalence at 3, 6, 9 and 1-year follow-ups
  Verified by saliva cotinine

SECONDARY OUTCOMES:
Cognitive and Affective Mechanisms of Treatment | Daily assessments completed throughout the day at random and scheduled times from baseline to 3 months
  E-diary use will collect daily cognitive and affective data from each participant in order to reveal mechanisms of treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: David Williams, PhD, Principal Investigator — Brown University
Locations (1):
- Public Health Building @ 121 South Main St, Providence, Rhode Island, United States

REFERENCES:
- [Derived] LaRowe LR, Dunsiger SI, Williams DM. Acute exercise-induced changes in motivation and behavioral expectation for quitting smoking as predictors of smoking behavior in women. Psychol Addict Behav. 2023 May;37(3):475-482. doi: 10.1037/adb0000901. Epub 2022 Dec 1. PMID 36455006